CLINICAL TRIAL: NCT00270491
Title: A Multicenter Randomized Phase II Study Evaluating Tolerance and Efficacy of Capecitabine 5/7 Days With Weekly Paclitaxel Versus the Recommended Treatment Plan of Weekly Paclitaxel-capecitabine, in Patients With Metastatic Breast Cancer.
Brief Title: Capecitabine Associated With Weekly Paclitaxel in Metastatic Breast Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAXEL
Record Dates: First submitted 2005-12-26; First posted 2005-12-28 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Breast Cancer; Neoplasm Metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Paclitaxel; Capecitabine

INTERVENTIONS:
Drug: Paclitaxel
Drug: Capecitabine

SUMMARY:
Tolerance and efficacy of administration of capecitabine 5 out of 7 days associated with weekly paclitaxel compared to the recommended treatment plan of weekly paclitaxel - capecitabine, in patients with metastatic breast cancer.

DETAILED DESCRIPTION:
The purpose of this study is to know if we can optimize in term of tolerance even of efficacy the plan of administration of weekly paclitaxel associated with capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Femal patient aged > 18 years
* Histologically proven breast adenocarcinoma
* HER2 negative receptors
* previously received first or second line chemotherapy for metastatic disease
* previously treated with anthracycline and/or docetaxel in adjuvant and/or as first or second line therapy
* presence of one or several evaluable metastatic lesion(s)
* presence of at least one target lesion not previously irradiated
* previously treated with hormonotherapy in adjuvant or in metastatic line (treatment will be ceased upon patient registration in the study)
* ECOG Performance status < 2
* adequate biological values
* patient who has clearly given her consent by signing on informed consent form prior to participation

Exclusion Criteria:

* patient previously treated with paclitaxel or capecitabine for metastatic breast cancer
* patient with only local metastatic disease (with the exception of axillary lymph nodes)
* active symptomatic brain metastasis
* patient with an history of significant cardiovascular impairment (congestive heart failure> NYHA grade II, unstable angina or myocardial infraction within the past six months or serious cardiac arrhythmia)
* peripheric neuropathy grade ≥ 2
* history of another malignancy within past 5 years that could confound diagnosis or staging of breast cancer (with the exception of in situ cacinoma of the cervix or adequately treated basel cell carcinoma of the skin)
* patient with any medical or psychiatric condition that, in the opinion of the Principal Investigator, would preclude her from participating in this study
* patient with a known allergy to one or several of the study compounds
* patients who may not be regularly available due to geographical, social or family reasons
* history of renal, hepatic or metabolic pathology that could preclude with metabolism or elimination of the study product
* deficiencies of the upper intestinal tract, malabsorption syndrome
* patient who is pregnant, breast-feeding or using inadequate contraception

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2005-12; Primary Completion 2009-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
tolerance of the patients in the both groups.

SECONDARY OUTCOMES:
- Response rates and duration of response.
- Haematological and non-haematological toxicities.
- Progression free survival.
- Overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Rémy LARGILLIER, Physician, Principal Investigator — Centre ANTOINE LACASSAGNE - NICE (FRANCE)
Locations (1):
- Hôpital HOTEL DIEU, Paris, France